CLINICAL TRIAL: NCT06056037
Title: Making Universal, Free-of-charge Antiretroviral Therapy Work for Sexual and Gender Minority Youth in Brazil
Brief Title: Making ART Work Among Brazilian Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: University of California, Los Angeles (Other); Oswaldo Cruz Foundation (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2103002951; R34MH126894 (NIH)
Record Dates: First submitted 2023-09-19; First posted 2023-09-28 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hiv; Adherence, Medication
Keywords: Brazil; sexual and gender minority; adolescents; HIV; Medication adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence; Coitus | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Pilot randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PIs nor the individual conducting outcome assessments will know the status of the participants' randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Making ART Work (Experimental): A culturally tailored, theoretically grounded social support intervention that includes receipt of daily text messages and provider-facilitated group adherence counseling (4 sessions)
  Interventions: Behavioral: Experimental: Making ART Work; Behavioral: Standard of Care
- Standard of Care (Active Comparator): Standard clinical care referrals and basic medication adherence education
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Experimental: Making ART Work — A culturally tailored, theoretically grounded provider-facilitated group-based social support intervention (4 sessions) that emphasizes a collective approach to ART adherence and includes establishing a common understanding of ART, identifying potential barriers to ART adherence with a focus on social and structural barriers (e.g., stigma, relationship influences, family support, economic stressors), developing practical strategies to increase self-esteem and self-efficacy to enhance ART adherence, and generating and maintaining peer norms and support for ART adherence within one's social group. These sessions will include SGM youth-specific video vignettes that address the social/contextual realities faced by SGM YLWH in Brazil. Lastly, the intervention includes daily SMS text messaging that serve as both reminders and cognitive cues to take medication as prescribed.
  Arms: Making ART Work
Behavioral: Standard of Care — Prior to randomization, all participants will meet briefly with a counselor to assess current needs for standard HIV primary care and referrals to social and/or health (including mental health) services. If participants do not have a primary HIV care provider, they will be linked to a provider at INI-Fiocruz or their preferred clinic, where they can access free HIV care through the no-cost universal access program of the Brazilian Public Health System. Additionally, the counselor will provide necessary referrals as needed, e.g., for social, general health and/or mental health services. Additionally, in order to provide a baseline level of standardized adherence information, all participants will receive a brief adherence educational session, which consists of a review of medications and recommended dosing, adherence expectations, toxicity expectations, and medication misperceptions.

SUMMARY:
This study seeks to develop and pilot test a theory-based, integrated technology and counseling intervention to improve ART adherence among sexual and gender minority (SGM) young people living with HIV (ages 18-24) in Rio de Janeiro, Brazil. The intervention aims to improve social support, self-efficacy for taking ART, and teach skills for problem-solving barriers to promote better adherence.

DETAILED DESCRIPTION:
Background. Sexual and gender minority (SGM) youth account for the largest number of incident HIV infections in Brazil. Although HIV can be managed with ongoing antiretroviral therapy (ART), exceptionally high levels of adherence are required. Brazil has implemented a comprehensive HIV treatment program with broad access to ART, but this program does not specifically address barriers to optimal ART adherence, particularly for SGM youth who experience many challenges taking their medication as prescribed. Overview. This application seeks to develop and pilot test a theory-based, integrated technology and counseling intervention to improve ART adherence among HIV infected SGM youth (ages 15-24) in Rio de Janeiro, Brazil. The intervention aims to improve social support, self-efficacy for taking ART, and teach skills for problem-solving barriers to promote better adherence. To inform the content, structure, and format of the proposed intervention, the MPIs recently conducted focus groups with SGM youth (N = 18) and key informant interviews (N = 7) with medical providers and staff at local HIV service organizations working closely with SGM youth in Rio de Janeiro. Across focus groups and key informant interviews there was universal agreement that an intervention should capitalize on and enhance social support structures among SGM youth, and address their specific concerns, especially as related to the individual (e.g., ART side effects, mood, substance use), social (e.g., HIV/SGM stigma), and structural (e.g., clinic hours, transportation challenges) barriers that they regularly face. Theoretical Model. The intervention is guided by Social Cognitive and Social Support Theories and is grounded in the social and contextual realities of SGM youth living with HIV in Brazil. Specifically, social support is emphasized and informational, problem-solving and cognitive-behavioral "steps" are addressed over 4-group adherence counseling sessions, which include short video vignettes that seek to normalize adherence challenges. In addition, daily tailored SMS text messages are delivered as part of the intervention to facilitate social-cognitive cues to take medications as prescribed. Research Plan. Phase 1: Refine and enhance participant acceptability of the intervention and resolve any issues with intervention delivery/implementation; this will be achieved by convening and obtaining feedback from our youth community advisory board throughout this phase and subsequent phases; and by conducting an open-phase pilot with up to 12 SGM youth, with post-intervention exit interviews, as well as obtaining feedback from our youth community advisory board throughout this and subsequent phases. Phase 2: Examine, in a pilot randomized controlled trial, the feasibility, acceptability and potential impact of the proposed intervention among approximately 72 SGM youth who will be equally randomized to the intervention or a standard of care control condition with standard of care. The outcomes are improved ART adherence, retention in care and viral load suppression. Study assessments will be conducted at baseline, 3- and 6-months.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 24 years of age
* assigned male sex at birth
* identify as a gay or bisexual man, or a transgender woman or another gender identity along the feminine spectrum
* self-report living with HIV, and verified by medical chart review,
* self-report currently taking or prescribed ART for > 3 months
* self-report missing 2 or more doses of ART medications in any given week in the past month OR not virally suppressed (i.e., >40 copies/mL in past 3 months; via national outpatient data [SISCEL] or plasma viral load testing)
* owns a cell phone or willing to use one as part of the study

Exclusion Criteria:

* unable to give informed consent due to cognitive limitation, severe mental/physical illness or intoxication
* unable to read and/or write to an extent that would limit their ability to comprehend the informed consent
* lived in the greater Rio de Janeiro area for < 3 months or planning to move outside the area within the next year

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility: number of participants who have at least one follow up visit | 6 months
  Retention rate
Feasibility: mean number of intervention sessions attended | 3 months
  Session attendance (in intervention arm)
Acceptability: mean score on the Client Satisfaction Questionnaire scale (CSQ-8) | 3 months
  CSQ-8
Medication adherence - proportion of participants with presence of tenofovir in urine using a point-of-care lateral flow immunoassay (LFA) method | 6 months
  Presence of tenofovir in urine using a point-of-care lateral flow immunoassay (LFA) method
Medication adherence - proportion who have received all ART prescriptions over the course of follow up according to pharmacy dispensing records (SICLOM national registry) | 6 months
  pharmacy dispensing records via the SICLOM database

SECONDARY OUTCOMES:
Plasma viral load - mean viral load as obtained through the SISCEL database (national registry) | 6 months
  verified via the SISCEL database
Retention in HIV care: proportion who have been in continuous care according to 1) at least 1 or more routine HIV visits, 3 months apart or more, (2) receiving 1 or more CD4 tests; and (3) receiving 1 or more viral load tests | 6 months
  verified using the SISCEL and SICLOM databases and medical records

CONTACTS AND LOCATIONS:
Overall Officials: Katie Biello, PhD, MPH, Principal Investigator — Brown University
Locations (1):
- Evandro Chagas National Institute of Infectious Diseases (INI) Oswaldo Cruz Foundation (FIOCRUZ), Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Raw data for additional analysis will be available to outside individuals through contacting the MPIs at two different times. The first will be after all of the baseline data is collected. We will institute a concept plan process where internal study staff first have the availability to write primary papers or give presentations on particular topics. After this, if outside individuals wish to analyze data, we will welcome this collaboration. A similar process will happen for outcome data; however this will not be possible until the publication and release of the outcome paper(s). The PI will store the data indefinitely and allow access for pooled data analysis projects, or projects for outside individuals. Information regarding the availability of data for analysis will be listed on the MPIs' web pages. Contact information for the PI will be listed in all manuscripts and publications as another means to access data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Raw data for additional analysis will be available to outside individuals through contacting the MPIs at two different times. The first will be after all of the baseline data is collected. We will institute a concept plan process where internal study staff first have the availability to write primary papers or give presentations on particular topics. After this, if outside individuals wish to analyze data, we will welcome this collaboration. A similar process will happen for outcome data; however this will not be possible until the publication and release of the outcome paper(s). The PI will store the data indefinitely and allow access for pooled data analysis projects, or projects for outside individuals.